CLINICAL TRIAL: NCT02742649
Title: A Phase 1B, Multicenter, Randomized, Double-masked, Controlled Study to Evaluate the Efficacy and Safety of a Fixed Combination Bimatoprost/Timolol Ocular Insert Compared to Its Individual Components With Crossover to Timolol 0.5% in Subjects With Open-angle Glaucoma (OAG) or Ocular Hypertension (OHT)
Brief Title: A Study to Evaluate Efficacy and Safety of a Fixed Combination Ocular Insert in Participants With Open-angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FSV5-FC-001
Record Dates: First submitted 2016-04-06; First posted 2016-04-19 (Estimated); Results first posted 2018-12-31 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost; Timolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fixed Combination (FC) Ocular Insert (Experimental): Washout plus Placebo Ocular Insert in each eye for 24 to 48 days, followed by one segment of bimatoprost and one segment of timolol maleate combined onto a single ocular insert in each eye for 70 days. Following a second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
  Interventions: Drug: Fixed Combination; Device: Placebo Segment; Drug: Timolol 0.5%
- Bimatoprost Ocular Insert (Experimental): Washout plus Placebo Ocular Insert in each eye for 24 to 48 days, followed by one segment of bimatoprost and one placebo segment (no drug product) combined onto a single ocular insert in each eye for 70 days. Following a second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
  Interventions: Drug: Bimatoprost; Device: Placebo Segment; Drug: Timolol 0.5%
- Timolol Ocular Insert (Experimental): Washout plus Placebo Ocular Insert in each eye for 24 to 48 days, followed by one segment of timolol and one placebo segment (no drug product) combined onto a single ocular insert in each eye for 70 days. Following a second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
  Interventions: Drug: Timolol; Device: Placebo Segment; Drug: Timolol 0.5%

INTERVENTIONS:
Drug: Fixed Combination — Continuous elution from the ocular insert.
  Other Names: Bimatoprost-Timolol combination
  Arms: Fixed Combination (FC) Ocular Insert
Drug: Bimatoprost — Continuous elution from the ocular insert. This is an active control arm.
  Other Names: Bimatoprost component only
  Arms: Bimatoprost Ocular Insert
Drug: Timolol — Continuous elution from the ocular insert. This is an active control arm.
  Other Names: Timolol component only
  Arms: Timolol Ocular Insert
Device: Placebo Segment — One segment of placebo (no drug product)
Drug: Timolol 0.5% — 0.5% timolol drops twice daily.

SUMMARY:
The purpose of this study is to determine if a combination of two drugs (bimatoprost and timolol) delivered to the surface of the eye over 10 weeks is better at lowering intraocular pressure (IOP) than either of the drugs delivered alone.

ELIGIBILITY:
Key Inclusion Criteria:

* Written informed consent
* At least 18 years of age
* Diagnosis in both eyes of either primary open-angle glaucoma (POAG) or ocular hypertension
* Best corrected-distance visual acuity score equivalent to 20/80 or better
* Stable visual field
* Central corneal thickness between 490 - 620 micrometers

Inclusion Criteria at the Randomization Visit:

* IOP for each eye is ≥ 23 mmHg at T=0hr, ≥ 20 mmHg at T=4hr and T=8hr.
* Inter-eye IOP difference of ≤ 5.0 mmHg at T=0hr, T=4hr and T=8hr.
* IOP for each eye is ≤ 30 mmHg at T=0hr, T=4hr and T=8hr.

Key Exclusion Criteria:

* Any known contraindication to prostaglandin analog (latanoprost, travoprost, bimatoprost, tafluprost) or timolol
* A cardiac or pulmonary condition that in the opinion of the Investigator would contraindicate the use of a topical beta-blocker
* Use of any agents known to have a substantial effect on IOP during planned study period (e.g. beta-blockers)
* Cup-to-disc ratio of greater than 0.8
* Significant risk of angle closure due to pupil dilation, defined as a Shaffer classification of less than Grade 2 based on gonioscopy
* Ocular, orbital, and/or eyelid surgery of any type within the past six (6) months from screening date
* Laser surgery for glaucoma / ocular hypertension on one (1) or both eyes within the last six (6) months
* Past history of any incisional surgery for glaucoma at any time
* Past history of corneal refractive surgery
* Corneal abnormalities that would interfere with accurate IOP readings with an applanation tonometer
* Current participation in an investigational drug or device study or participation in such a study within 7 days of Screening
* Inability to adequately evaluate the retina
* Subjects who will require contact lens use during the study period.
* Subjects who currently have punctal occlusion
* Pregnant, lactating or of child-bearing potential and not using a medically acceptable form of birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-04-30 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chen, PhD, Study Director — Allergan
Locations (1):
- Clinica de Ojos Orillac - Calvo, Panama City, Panama

RESULTS

PARTICIPANT FLOW:
Groups:
- Washout + Placebo Ocular Insert: During the washout period, participants wore a placebo insert in each eye serving as a trial-wear period for 24 to 48 days.
- Fixed Combination (FC) Ocular Insert: Following washout period, one segment of bimatoprost and one segment of timolol maleate were combined in an ocular ring and inserted in each eye for 70 days, followed by a second washout period from Day 71 to 98.
- Bimatoprost Ocular Insert: Following washout period, one segment of bimatoprost and one placebo segment were combined in an ocular ring and inserted in each eye for 70 days followed by a second washout period from Day 71 to 98.
- Timolol Ocular Insert: Following washout period, one segment of timolol and one placebo segment were combined into an ocular ring and inserted in each eye for 70 days, followed by a second washout period from Day 71 to 98.
- Timolol 0.5% Ophthalmic Drops: Following a second washout period, timolol drops, 0.5% solution twice daily in each eye from Day 99 to 112.
Period: Pre-Randomization Washout Period
Arm/Group | Washout + Placebo Ocular Insert | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert | Timolol 0.5% Ophthalmic Drops
Started | 55 | 0 | 0 | 0 | 0
Completed | 50 | 0 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0 | 0
Not completed — Washout/Randomization Failure | 5 | 0 | 0 | 0 | 0
Period: Double-Blind Treatment Period
Arm/Group | Washout + Placebo Ocular Insert | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert | Timolol 0.5% Ophthalmic Drops
Started | 0 | 17 | 17 | 16 | 0
Completed | 0 | 16 | 17 | 16 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Period: Open-Label Period
Arm/Group | Washout + Placebo Ocular Insert | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert | Timolol 0.5% Ophthalmic Drops
Started | 0 | 0 | 0 | 0 | 49
Completed | 0 | 0 | 0 | 0 | 48
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) included all participants who were randomized, treated and returned for at least one (1) regularly scheduled post-treatment visit. Participants were analyzed in the treatment group to which they were randomized (Double Blind Treatment Period).
Groups:
- Fixed Combination (FC) Ocular Inset: Following washout period, one segment of bimatoprost and one segment of timolol maleate were combined in an ocular ring and inserted in each eye for 70 days, followed by a second washout period from Day 71 to 98. Following the second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
- Bimatoprost Ocular Insert: Following washout period, one segment of bimatoprost and one placebo segment were combined in an ocular ring and inserted in each eye for 70 days followed by a second washout period from Day 71 to 98. Following the second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
- Timolol Ocular Insert: Following washout period, one segment of timolol and one placebo segment were combined into an ocular ring and inserted in each eye for 70 days, followed by a second washout period from Day 71 to 98. Following the second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
- Total: Total of all reporting groups
Arm/Group | Fixed Combination (FC) Ocular Inset | Bimatoprost Ocular Insert | Timolol Ocular Insert | Total
Number analyzed (Participants) | 17 | 17 | 16 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.24 (12.94) | 68.94 (5.75) | 67.56 (9.27) | 67.92 (9.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 11 | 36
  Male | 3 | 6 | 5 | 14
Intraocular Pressure (IOP) [Mean (Standard Deviation); unit: mm Hg] — IOP is a measurement of the fluid pressure inside the eye. IOP was measured at the following three time points: 8 am (T=0 hour), 12 pm (T=4 hour) and 4 pm (T=8 hour). The IOP measured in the two eyes was averaged to compute a single IOP value for each timepoint.
  mm Hg
    Randomization (T=0 hour) | 24.34 (2.06) | 24.30 (1.89) | 24.18 (1.78) | 24.27 (1.88)
    Randomization (T=4 hour) | 22.98 (2.92) | 22.93 (3.06) | 23.33 (2.77) | 23.07 (2.87)
    Randomization (T=8 hour) | 22.44 (2.57) | 22.90 (3.13) | 23.03 (2.70) | 22.78 (2.77)

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure (IOP) on Day 8
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured at the following three time points: 8 am (T=0 hour), 12 pm (T=4 hour) and 4 pm (T=8 hour). The IOP measured in the two eyes was averaged to compute a single IOP value for each timepoint.
Time Frame: Day 8
Population: FAS included all participants who were randomized, treated and returned for at least one (1) regularly scheduled post-treatment visit. Participants were analyzed in the treatment group to which they were randomized (Double Blind Treatment Period).
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 17 | 17 | 16
mm Hg
  Day 8 (T=0 hour) | 17.83 (3.39) | 19.15 (2.62) | 19.59 (4.68)
  Day 8 (T=4 hour) | 17.51 (3.18) | 18.96 (4.14) | 19.88 (5.42)
  Day 8 (T=8 hour) | 17.05 (3.32) | 17.84 (4.00) | 19.66 (4.54)

2. Primary Outcome: IOP on Day 16
Description: as for outcome 1
Time Frame: Day 16
Population: FAS included all participants who were randomized, treated and returned for at least one (1) regularly scheduled post-treatment visit. Participants were analyzed in the treatment group to which they were randomized (Double Blind Treatment Period). Number analyzed is the number of participants with data at the given time-point.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 15 | 17 | 16
mm Hg
  Day 16 (T=0 hour) | 18.29 (3.86) | 18.08 (3.98) | 20.81 (5.22)
  Day 16 (T=4 hour) | 17.95 (3.10) | 18.64 (4.17) | 21.08 (5.46)
  Day 16 (T=8 hour) | 17.21 (4.14) | 18.54 (3.73) | 19.43 (3.77)

3. Primary Outcome: IOP on Day 28
Description: as for outcome 1
Time Frame: Day 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 16 | 17 | 16
mm Hg
  Day 28 (T=0 hour) | 18.03 (4.21) | 18.44 (4.23) | 19.75 (4.80)
  Day 28 (T=4 hour) | 18.54 (3.50) | 19.59 (3.70) | 20.09 (4.67)
  Day 28 (T=8 hour) | 17.26 (2.60) | 18.77 (4.13) | 19.20 (3.60)

4. Primary Outcome: IOP on Day 49
Description: as for outcome 1
Time Frame: Day 49
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 15 | 17 | 16
mm Hg
  Day 49 (T=0 hour) | 18.55 (4.05) | 18.88 (4.52) | 18.63 (3.89)
  Day 49 (T=4 hour) | 17.77 (4.02) | 19.35 (3.51) | 19.67 (3.54)
  Day 49 (T=8 hour) | 17.23 (4.53) | 18.48 (3.57) | 19.13 (2.40)

5. Primary Outcome: IOP on Day 70
Description: as for outcome 1
Time Frame: Day 70
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Groups:
- Fixed Combination (FC) Ocular Insert: Following washout period, one segment of bimatoprost and one segment of timolol maleate were combined in an ocular ring and inserted in each eye for 70 days, followed by a second washout period from Day 71 to 98. Following the second washout period, 0.5% timolol drops twice daily in each eye from Day 99 to 112.
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 16 | 17 | 16
mm Hg
  Day 70 (T=0 hour) | 17.60 (2.94) | 17.78 (2.58) | 17.79 (4.36)
  Day 70 (T=4 hour) | 18.09 (3.73) | 18.71 (3.59) | 18.48 (4.23)
  Day 70 (T=8 hour) | 17.14 (2.64) | 18.61 (4.07) | 18.78 (4.13)

6. Secondary Outcome: Number of Participants With Ocular and Non-Ocular Adverse Events
Description: An adverse event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Reported here is the number of participants with adverse events related to the eye as well as number of participants with all other adverse events.
Time Frame: From Randomization (Day 0) to Day 70
Population: Safety population set included all randomized participants who had an ocular insert placed at the Randomization Visit. In this analysis set, participants were analyzed according to the treatment received during each study treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 17 | 17 | 16
Participants
  Ocular | 13 | 14 | 10
  Non-Ocular | 11 | 10 | 5

7. Secondary Outcome: IOP During Open Label Period
Description: IOP is a measurement of the fluid pressure inside the eye. IOP was measured at the following three time points: 8 am (T=0 hour), 12 pm (T=4 hour) and 4 pm (T=8 hour) at the start (Day 98) and end (Day 112) of the Open Label Period during which participants were treated with timolol 0.5% ophthalmic solution twice daily. The IOP measured in the two eyes was averaged to compute a single IOP value for each timepoint.
Time Frame: Day 98, Day 112
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Fixed Combination (FC) Ocular Insert | Bimatoprost Ocular Insert | Timolol Ocular Insert
Number analyzed (Participants) | 17 | 17 | 16
mm Hg
  Day 98 (T=0 hour): number analyzed (Participants) | 16 | 17 | 16
  Day 98 (T=0 hour) | 22.61 (2.41) | 22.69 (3.06) | 23.24 (3.54)
  Day 98 (T=4 hour): number analyzed (Participants) | 16 | 17 | 16
  Day 98 (T=4 hour) | 21.67 (2.42) | 22.38 (3.16) | 22.99 (4.25)
  Day 98 (T=8 hour): number analyzed (Participants) | 16 | 17 | 16
  Day 98 (T=8 hour) | 20.74 (1.65) | 22.88 (3.89) | 22.63 (3.92)
  Day 112 (T=0 hour): number analyzed (Participants) | 16 | 17 | 15
  Day 112 (T=0 hour) | 19.21 (3.59) | 20.65 (3.90) | 19.71 (1.59)
  Day 112 (T=4 hour): number analyzed (Participants) | 16 | 17 | 15
  Day 112 (T=4 hour) | 17.62 (3.41) | 18.52 (3.97) | 18.75 (4.26)
  Day 112 (T=8 hour): number analyzed (Participants) | 16 | 17 | 15
  Day 112 (T=8 hour) | 17.51 (3.98) | 18.43 (4.45) | 18.19 (3.69)

ADVERSE EVENTS:
Time Frame: Randomization (Day 0) to the end of the study (Day 112)
Arm/Group | Fixed Combination (FC) Ocular Inset | Bimatoprost Ocular Insert | Timolol Ocular Insert
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 2/17 | 1/17 | 0/16
Other Adverse Events (participants affected / at risk) | 16/17 | 16/17 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Combination (FC) Ocular Inset (N=17) | Bimatoprost Ocular Insert (N=17) | Timolol Ocular Insert (N=16)
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0 — This was a planned procedure.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fixed Combination (FC) Ocular Inset (N=17) | Bimatoprost Ocular Insert (N=17) | Timolol Ocular Insert (N=16)
Eye discharge (Eye disorders) | 5 | 5 | 5
Conjunctival disorder (Eye disorders) | 4 | 2 | 5
Eye irritation (Eye disorders) | 5 | 4 | 2
Conjunctival hyperaemia (Eye disorders) | 5 | 2 | 1
Ocular discomfort (Eye disorders) | 4 | 3 | 1
Conjunctivitis (Eye disorders) | 3 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Punctate Keratitis (Eye disorders) | 3 | 1 | 1
Vision Blurred (Eye disorders) | 2 | 2 | 2
Eyelid Oedema (Eye disorders) | 0 | 2 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 7 | 2
Headache (Nervous system disorders) | 3 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Keratitis (Eye disorders) | 2 | 1 | 1
Foreign body sensation in eyes (Eye disorders) | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0 | 1
Dry eye (Eye disorders) | 0 | 1 | 0
Erythema of eyelid (Eye disorders) | 0 | 0 | 1
Lagophthalmos (Eye disorders) | 1 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0
Retinal artery occlusion (Eye disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No presentation or publication of Institution's data relating to the Trial may occur until after the Trial has been completed at all sites. If Investigator desires to present or publish, investigator must submit any and all manuscripts, posters, abstracts, or other intended publications (hereinafter collectively referred to as "manuscripts") to Sponsor at least sixty (60) days prior to the actual submission of such manuscript(s) for publication.